CLINICAL TRIAL: NCT03105011
Title: Utilizing Off-the-shelf Technology to Improve Diabetes Management in a Rural Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Morgan Carlile, Medical Student, University of Missouri-Columbia
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007269C
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EpxDiabetes software (Experimental): Subjects will interact daily with a commercially available telemedicine product, Epharmix Diabetes (EpxDiabetes).
  Interventions: Behavioral: EpxDiabetes software

INTERVENTIONS:
Behavioral: EpxDiabetes software — Subjects will interact daily with a commercially available telemedicine product, Epharmix Diabetes (EpxDiabetes). They will each undergo a baseline blood draw to establish the control HgbA1C associated with standard of care. Three months later they will undergo an experimental blood draw to establish the HgbA1C associated with the use of EpxDiabetes. Between those procedures, the patient will interact with the intervention daily.
  Other Names: Epharmix Diabetes

SUMMARY:
This study is designed to see if rural patients with type II diabetes interacting with their clinic staff by providing daily updates of blood glucose levels will improve glucose control.

DETAILED DESCRIPTION:
Hypothesis: Intervening in a rural primary care population with a clinically validated telehealth tool (Epharmix Diabetes) that algorithmically triages patients and facilitates patient-provider communication will result in a statistically significant improvement in the indicators of diabetes control.

Study Design

* Study Type: Experimental, non-controlled crossover study (intervention vs. standard of care for clinic)
* Primary aim: decrease average self-tested pre-prandial blood glucose level and HgbA1C
* Secondary aim: decreased number of disease-related emergency room (ER) visits, decreased number of self-reported blood glucose measurements outside of goal
* Duration: 3 months + 1 month enrollment period
* Safety: Protocol will be under direction of University of Missouri Institutional Review Board (IRB). All patients will be referred to emergency department if unsafe blood glucose levels are reported. All information is encrypted and HIPAA compliant.
* Sample Size: Clinic flow analysis estimates 61 patients eligible for study (5 providers, assuming 30% of eligible patients who meet inclusion criteria during 4-week enrollment period interested), with 50 patients likely to stay in study (80% retention rate).
* Power analysis: Based on pilot data and assuming an alpha error = 0.05, this study will have have greater than 80% statistical power of detecting differences in populations using only 20 patients with a minimum detectable effect size (decrease in HgbA1C) of 0.7%

Methodology

* The investigator will supply family practice clinics at Mercy with a one-page summary and advertisement of the intervention. At some point during a clinical encounter with a patient with an existing or new diagnosis of diabetes, providers will invite the patient to participate in this Community Integration Project. Providers will maintain a list of patients interested in the study with corresponding phone numbers and the investigator will regularly add patients to the study.
* Over a 3-month study period, patients will interact with the telehealth system twice a day, entering blood glucose levels when prompted. As recommended by physicians at Mercy, the investigator will message the physicians once a week with a digest of their patients at risk through the existing electronic medical record (EMR) inbox to more easily integrate with existing clinic flow.
* HgbA1c will be measured prior to starting intervention and will be measured within 7 days of completing intervention.
* Providers will be notified by the system when patients are triaged to be "high risk," that is, out of a pre-selected range of self-reported blood glucose levels. Providers can then be automatically connected with these patients to titrate blood glucose control.
* At the conclusion of study, new average self-reported blood glucose responses will be compared against those averages prior to intervention and to clinic averages for patients with diabetes. Additionally, HgbA1C levels will be compared pre and post -intervention.
* Results will be analyzed and conclusions will be presented to participating stakeholders in a poster session.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years of age
2. Gender: Any gender
3. Language: patients must use English as primary language
4. Patient must be ambulatory patients at Mercy Family Practice Clinic in Rolla, Missouri
5. Patient must have access to touch tone telephone or mobile phone with texting capability
6. Patient must have documented type 2 diabetes mellitus with a treatment plan that includes measuring pre-prandial blood glucose levels each morning.
7. HgbA1c between 7 and 9%

Exclusion Criteria:

* Patients that are identified by clinic staff who have demonstrated noncompliance
* Lack of access to mobile or landline telephone
* Hospitalized patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Absolute change in laboratory-measured HgbA1C | Baseline, 3 months
  Patients will undergo two diagnostic blood collections to measure baseline and final HgbA1C.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan A Carlile, Principal Investigator — University of Missouri-Columbia; Uzma Khan, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No